CLINICAL TRIAL: NCT00910637
Title: Multicenter, Open-label, Uncontrolled Study to Investigate the Efficacy and Safety of the Transdermal Contraceptive Patch Containing 0.55 mg Ethinyl Estradiol and 2.1 mg Gestodene in a 21-day Regimen for 13 Cycles in 1650 Healthy Female Subjects
Brief Title: Study Investigating the Efficacy and Safety of a Contraceptive Patch for 13 Cycles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 91555; 310802 (Other: Company internal)
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Contraception
Keywords: Pregnancy prevention; Female contraception; Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Gestodene/EE Patch (BAY86-5016)

INTERVENTIONS:
Drug: Gestodene/EE Patch (BAY86-5016) — 55 mg ethinyl estradiol & 2.1 mg gestodene, 21 days for 13 cycles

SUMMARY:
This study is examining a birth control patch for 13 cycles (1 year).

ELIGIBILITY:
Inclusion Criteria:

* Requiring contraception
* Normal cervical smear
* Maximum age for smokers is 35
* History of regular cyclic menstrual periods

Exclusion Criteria:

* Pregnancy or lactation
* Significant skin reaction to transdermal preparations or sensitivity to surgical / medical tape
* Any disease that may worsen under hormonal treatment (cardiovascular, liver, metabolic)
* Use of other contraceptive methods than study medication

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1502 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2010-12-13 (Actual); Study Completion 2010-12-13 (Actual)

PRIMARY OUTCOMES:
Occurrence of pregnancy (yes/no) while on treatment | 13 treatment cycles each consisting of 28 days and follow-up period of 14 days

SECONDARY OUTCOMES:
Vital signs | 13 treatment cycles each consisting of 28 days
Physical and gynecological examinations | 13 treatment cycles each consisting of 28 days
Laboratory assessments | 13 treatment cycles each consisting of 28 days
Adverse events (AE monitoring) | 13 treatment cycles each consisting of 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (60):
- United States (60):
  - Birmingham, Alabama
  - Glendale, Arizona
  - Precision Trials, Phoenix, Arizona
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Carmichael, California
  - Pacific Palisades, California
  - Paramount, California
  - Genesis Center for Clinical Research, San Diego, California
  - San Diego, California
  - Santa Ana, California
  - Torrance, California
  - Denver, Colorado
  - Littleton, Colorado
  - New London, Connecticut
  - Visions Clinical Research, Boynton Beach, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Meridien Research, St. Petersburg, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Roswell, Georgia
  - Research Associates, Boise, Idaho
  - Rosemark Women Care Specialist, Idaho Falls, Idaho
  - Chicago, Illinois
  - Newburgh, Indiana
  - South Bend, Indiana
  - Marrero, Louisiana
  - Boston, Massachusetts
  - Chaska, Minnesota
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Office of Dr. R. Garn Mabey, MD, Las Vegas, Nevada
  - Lawrenceville, New Jersey
  - Moorestown, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - York Clinical Consulting, Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Warwick, Rhode Island
  - Columbia, South Carolina
  - Mt. Pleasant, South Carolina
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Women's Care Center, PLC, Memphis, Tennessee
  - Nashville, Tennessee
  - Corpus Christi, Texas
  - Practice Research Organization, Dallas, Texas
  - Advances in Health, inc., Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - Norfolk, Virginia
  - Women's Clinical Research Center, Seattle, Washington